CLINICAL TRIAL: NCT02573038
Title: Phase II Study Evaluating the Efficacy of Aflibercept for the Treatment of Choroidal Neovascularization in Angioid Streaks in Young Patients.
Brief Title: Phase II Study Evaluating the Efficacy of Aflibercept for the Treatment of Choroidal Neovascularization in Angioid Streaks in Young Patients (ASTRID).
Acronym: ASTRID
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014.878; 2014-003661-18 (EudraCT Number)
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Choroidal Neovascularization in Angioid Streaks
Keywords: Aflibercept; choroidal neovascularization; angioid streaks; young patient
MeSH Terms: conditions — Choroidal Neovascularization; Angioid Streaks | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aflibercept (Experimental): Intravitreal injection of aflibercept (EYLEA) / 2mg
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — The patients are followed on a monthly basis until 52 weeks. Intravitreal injections of aflibercept at a dosage of 2 mg are initiated at inclusion (mandatory injection) followed by mandatory injections at week 4, week 8, week 20, week 32 and week 44. During the other visits, an injection can be performed in case of CNV activity (PRN regimen).Therefore, each patient receives between 6 and 13 injections in the whole study.

SUMMARY:
Angioid streaks are rare lesions associated to retinal pigment epithelium degenerations.

They can be caused by general diseases as pseudoxanthoma elasticum, Paget's disease or drepanocytosis. Choroidal neovascularization (CNV) represents the most frequent complication for those patients. It leads to a rapid and important loss of visual acuity. CNV in angioid streaks represent the fourth leading cause of CNV in young patients.

CNV in angioid streaks is treated at the moment with off-label anti-VEGF (Vascular Endothelial Growth Factor) therapy and could also benefit from aflibercept (EYLEA), a new anti-VEGF currently indicated in AMD. Case reports suggest that such patients would not need as many injections as in AMD.

ASTRID is an open-label, single arm, prospective, multicenter, phase II study. The main objective is to demonstrate the effectiveness in clinical terms after 52 weeks of treatment with aflibercept on the visual acuity of patients affected by CNV in angioid streaks. A specific dosage regimen is designed to achieve maximum efficiency. The patients are followed on a monthly basis until 52 weeks. Six injections are mandatory, the other ones are injected only in case of active CNV.

ELIGIBILITY:
Inclusion Criteria:

* 18 < Age < 50 years old
* Patient who give voluntary signed informed consent
* Patient affiliated with the French universal health care system or similar
* Patient with CNV in angioid streaks, whatever caused the angioid streaks, with active primary subfoveal, retrofoveal or juxtafoveal lesions that affect the fovea as evidenced by angiography (fluorescein and/or indocyanine green) and/or SD-OCT in the studied eye
* Patient willing, committed and able to return for all clinic visits and complete all study-related procedures

Exclusion Criteria:

* Pregnant women
* Sexually active men or women of childbearing potential who are unwilling to practice adequate contraception during the study
* Patient who is protected adults according to the terms of the law (French public health laws)
* Involvement in another clinical trial (studied eye and/or the other eye)
* Patient with non-angioid streaks CNV, especially:

  * AMD
  * High myopia defined as refraction ≥ - 6 diopters
* Other curative treatment of CNV in angioid streaks in the studied eye during the last 3 months before the first intravitreal injection: anti-VEGF therapy, juxta- or extra-foveal macular laser, photodynamic therapy, surgery, external radiotherapy, transpupillary thermotherapy ...
* Medical history of retrofoveal focal macular laser photocoagulation in the studied eye
* Subretinal hemorrhage reaching the fovea center or with a size > 50% of the lesion area
* Fibrosis or retrofoveal retinal atrophy in the studied eye
* Retinal pigment epithelial tear reaching the macula in the studied eye
* Medical history of intravitreal medical device in the studied eye
* Medical history of auto-immune or idiopathic uveitis
* Proved diabetic retinopathy
* Intra-ocular pressure ≥ 25 mmHg despite two topical hypotonic treatments
* Aphakia or lack of lens capsule (not removed by YAG laser) in the studied eye
* Arterial hypertension that is not controlled by an appropriate treatment and defined by one measure of systolic blood pressure > 180mmHG or 2 consecutive measures > 160mmHg, or by a diastolic blood pressure > 100mmHg
* Antecedents of cerebrovascular disease or myocardial infarction during the last 6 months before inclusion (J1)
* Antecedents of any pathology, metabolic disease, or any serious suspicion of disease during the clinical or laboratory exam that would contraindicate the use of the product, could affect the interpretation of the study results or lead to major risks of complication for the subject
* Renal insufficiency requiring dialysis or renal transplantation
* Previous (less than a year) or actual treatment with systemic administration of anti-VEGF therapy
* Known hypersensitivity to aflibercept, or another drug composite of the medicinal product used; allergy to fluorescein, indocyanine green, anaesthetic eye drops
* Active or suspected ocular or peri-ocular infection
* Active severe intraocular inflammation
* Medical history of intra-ocular surgery within 28 days before the first injection in the studied eye
* Any illness or ocular condition that would require an intra-ocular surgery in the studied eye within 12 months after the inclusion
* Follow up not possible during 12 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Mean change in best corrected visual acuity (BCVA) from baseline to 52 weeks in patients with choroidal neovascularization in angioid streaks treated with Aflibercept | 52 weeks
  Change in BCVA number of letters gained or lost between baseline and 52 weeks. BCVA is measured on the scale Early Treatment Diabetic Retinopathy Study (ETDRS) at an initial distance of 4 meters.

SECONDARY OUTCOMES:
Mean change in BCVA from baseline to 24 weeks | 24 weeks
  Mean change in BCVA expressed as number of letters gained or lost measured with ETDRS scale from baseline to week 24
Percentage of patients who lost fewer than 15 letters of BCVA from baseline to 24 weeks. | 24 weeks
  percentage of the patients who lost fewer than 15 letters of BCVA measured with ETDRS scale from baseline to week 24.
Percentage of patients who lost fewer than 15 letters of BCVA from baseline to 52 weeks | 52 weeks
  Percentage of the patients who lost fewer than 15 letters of BCVA measured with ETDRS scale from baseline to week 52.
number of injections per patient for 52 weeks | 52 weeks
Average change in central retinal thickness (CRT) between baseline and 24 weeks | 24 weeks
  Average change in central retinal thickness (CRT) in micrometers measured with Spectral domain Optical Coherence Tomography (SD-OCT) from baseline to week 24
Average change in central retinal thickness (CRT) between baseline and 52 weeks | 52 weeks
  Average change in central retinal thickness (CRT) in micrometers measured with Spectral domain Optical Coherence Tomography (SD-OCT) from baseline to week 52
Mean change in neovascular lesion size between baseline and 52 weeks. | 52 weeks
  change in neovascular lesion size measured with fluorescein and/or indocyanine green angiography from baseline to week 52
Mean change in neovascular lesion morphology between baseline and 52 weeks. | 52 weeks
  Mean change in neovascular lesion morphology measured with fluorescein and/or indocyanine green angiography from baseline to week 52
Side-effects observed during the study | 52 weeks